CLINICAL TRIAL: NCT03085277
Title: Bovine Colostrum Versus Preterm Formula as the First Supplemental Nutrition for Very Preterm Infants, a Randomized, Controlled Trial
Brief Title: Bovine Colostrum for Preterm Newborns
Acronym: PreColos-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Per Torp Sangild (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other); Maternal and Child Health Hospital of Foshan (Other); Shenzhen People's Hospital (Other); Shenzhen Luohu Maternal and Child Health Hospital (Unknown); University of Chinese Academy of Sciences - Shenzhen Hospital (Unknown); Longgang District People's Hospital of Shenzhen (Other); Shenzhen Nanshan Maternity and Child Healthcare Hospital (Unknown); Dongguan Women and Children's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Per Torp Sangild, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Precolos-RCT
Record Dates: First submitted 2017-03-14; First posted 2017-03-21 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Enteral Feeding Intolerance; Necrotizing Enterocolitis; Late-Onset Neonatal Sepsis
Keywords: Bovine colostrum; Preterm formula; Very preterm infants; Enteral feeding
MeSH Terms: conditions — Enterocolitis, Necrotizing; Neonatal Sepsis

STUDY DESIGN:
Intervention Model Description: When a preterm infant is delivered at these hospitals or transferred from other hospitals on the day of birth, responsible neonatologists/PIs/co-PIs will evaluate the infant for its eligibility. If the infant fulfills the recruitment criteria, parent(s) are informed and explained about the study and asked for permission to recruit their babies. After confirmed consent, the infant will be, per hospital, randomized to two groups in a 1:1 ratio. Infants should be recruited and randomized as soon as possible after birth and no later than 48 h. The first supplemental enteral feeding (PF or BC) can be given as soon as the infants are randomized. Randomization will be stratified by birth weight < 1000 g, birth weight ≥ 1000 g, and randomly permuted blocks of size 4 and 6 will be used. A random sequence list will be generated by computer software for each hospital and a corresponding sequence number can only be checked to see allocation after informed consent is given and the baby is enrolled.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preterm Formula (Active Comparator): MM is always the first priority, when available. When MM is not available, or the available amounts do not fulfill the needs, infants in this group will receive preterm formula, as the supplementary diets following the standard feeding guidelines in the participating hospitals.
  Interventions: Dietary Supplement: Preterm Formula
- Bovine Colostrum (Experimental): MM is always the first priority, when available. When MM is not available, or the available amounts do not fulfill the needs, infants in this group will receive Bovine Colostrum (BC), as the supplementary diets. BC feeding follows the same guideline as the control group in terms of initiation time (within 24-48h of age) and volume (5-10 ml/kg) and advancing rate (5-20 ml/kg/d). BC intervention should not exceed postnatal day 14.
  Interventions: Dietary Supplement: Bovine Colostrum

INTERVENTIONS:
Dietary Supplement: Bovine Colostrum — Bovine colostrum (BC) is the first milk from cows after birth and we suggest that BC may be used to supplement MM, instead of infant formula or DM. BC is a rich source of protein (up to 150 g/L) and bioactive components, including lactoferrin, lysozyme, lactoperoxidase, immunoglobulins, and various growth factors, such as, IGF-I and -II, EGFs, and TGF-β. BC has repeatedly been shown to have beneficial effects in a well-established piglet model of preterm infants, using various feeding regimens, including a gradual regimen that would mimic enteral feeding for preterm infants without access to MM during the first week.
  Arms: Bovine Colostrum
Dietary Supplement: Preterm Formula — Preterm formula is a type of infant formula designed for preterm infants. It is used when mother's own milk is not available or not in sufficient amount as the enteral feeding for preterm infants in hospitals that do not have donor human milk.
  Arms: Preterm Formula

SUMMARY:
Feeding intolerance is a common problem in very preterm infants due to their immature digestive system. This intolerance extends the time to full enteral feeding and thereby also prolongs the time on parenteral nutrition (PN). Prolonged time to full enteral feeding may predispose these infants to a higher risk of growth retardation, infections and organ dysfunctions (e.g. liver, brain). Mother's own milk (MM) is considered the optimal nutrition for preterm infants and is superior to infant formula (including preterm formula, PF) in stimulating gut maturation, feeding tolerance, resistance against necrotizing enterocolitis (NEC) and late-onset sepsis (LOS), and long-term neurodevelopmental outcomes. However, MM is often absent, or not available in sufficient amounts, during the first days or weeks after preterm delivery. Human donor milk (DM) is probably a better supplement to MM than PF, but DM is not available for all hospitals. To supplement insufficient MM during the early neonatal period in hospital settings with no access to donor milk, we suggest that bovine colostrum (BC) may be used instead of PF for very preterm infants during early life. BC, the first milk from cows after birth, is a rich source of protein and bioactive components, including lactoferrin, lysozyme, lactoperoxidase, immunoglobulins, and various growth factors, such as IGF-I and -II, EGFs, and TGF-β. BC has repeatedly been shown to improve gut maturation and NEC/LOS resistance in a well-established piglet model of preterm infants. We suggest a randomized, controlled trial to investigate the effects of BC vs. PF, supplemented to MM during the first 2 weeks, on the time to full enteral feeding in very preterm infants.

DETAILED DESCRIPTION:
The Precolos-RCT is a multicenter, two-arm, unblinded, randomized, controlled trial. Infants are randomized to an intervention group which receives BC and a control group which receives PF. In detail, MM is always the first priority, when available. When MM is not available, or the available amounts do not fulfill the needs, infants in BC group will receive BC and control infants will receive PF, as the supplementary diets. Feeding should be initiated within 24-48 h after birth following a pre-defined nutritional guideline. BC intervention should not exceed postnatal day 14. After the intervention period, the participants in both groups will receive standard feeding which is the available MM with or without supplemental preterm infant formula. Infants will be followed until discharge home or reach a postconceptional age of 37 weeks, whichever comes first (discharge home/37 wks).

In general, parenteral and enteral nutrition should be given according to the following description:

Parenteral and enteral nutrition will be given according to the targeted daily fluid, energy, and protein levels suggested by ESPGHAN and CSPEN. Enteral nutrition should be given according to the feeding guideline and PN is used to ensure the targeted protein, energy, and lipid intake when enteral feeding is insufficient to provide fluid and nutrition. Participating hospitals should try their best to assist mothers in expressing their colostrum and milk and giving mother's colostrum as the first feeds. Enteral feeding should be given as soon as possible within 24h of life after randomization for infants with BW > 750g. For infants with BW ≤ 750 g, first feeding should be given within 24 h if mother's colostrum is available. Otherwise, first feeding should wait until day 2 for mothers to express their own colostrum. Mother's colostrum and MM is given as much as available, and when it is not available or in an insufficient amount, BC or PF is used during the intervention period to supplement the lacking volume. Infants should receive an initial feeding volume of 5-10 ml/kg/d and the volume should increase by 5-20 ml/kg/d until 150-160 ml/kg/d depending on their BW. The advancing rate of feeding should follow the suggested pace but also be adjusted according to the tolerability of the infants. If feeding intolerance occurs, feeding should be at a flat rate or be withheld according to predefined criteria in 'parenteral and enteral nutrition SOP'. If infants can tolerate more, feeding can be increased faster. Since total protein intake should be within 4-4.5 g/kg/d according to the ESPGHAN guideline25, the maximal daily volume of BC should be calculated based on the available volume of MM and protein levels in MM and BC. The protein supply from MM is calculated assuming a protein content of 1.5 g/100 mL27 (during the first 14 days) and the protein supply from colostrum is 8 g/100 mL (may adjust to changes according to the product specification of the batch in use when the difference is bigger than 5%). At the end of the intervention period, the enteral feeding in the intervention group will be gradually transferred to standard feeding (MM with supplemental PF when needed). Participants in the control group will keep receiving standard feeding after the intervention period. However, if a participant reaches term during their hospital stay, PF may be changed to term formulas according to local guidelines. The participating hospitals use four types of PF with similar nutrients composition and will remain the same throughout the study.

Although in the intervention group, infants should receive supplemental BC instead of PF during the intervention period, there is a possibility that PF and BC are simultaneously used as the supplemental diets. For example, when a participant in the intervention group can tolerate a higher EN volume than the available volume of MM plus the maximum daily volume of BC (due to max protein limitation), PF needs to be given to fulfill the total EN volume. Importantly, the volume of each milk diet will need to be adjusted according to the maximal protein intake of 4-4.5 g/kg/d. When BC intake has reached the maximal volume due to protein limitation but fluid requirement still needs to be fulfilled by PN, the PN should be given with an amino acid level of 0.5 g/kg/d （other nutrients are provided accordingly）and BC volume should be reduced by 6.25 ml/kg/d. A detailed guideline for parenteral and enteral nutrition is described in an SOP: 'Parenteral and enteral nutrition SOP'.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with gestational age between 26+0 and 31+6 weeks
* Delivered at participating hospitals or transferred from other hospitals within 24 h of age
* Signed parental consent

Exclusion Criteria:

* Major congenital anomalies or birth defects
* Congenital infection defined as suspected TORCHES infections: Toxoplasmosis, Rubella, CMV, Herpes, Hepatitis, Coxcackie, Syphilis, Varicella Zoster, HIV, Parvo B19
* Perinatal asphyxia with blood pH < 7.0 (umbilical or first neonatal)
* Extremely small for gestational age (birth weight z-score ≤ - 3)
* No realistic hope of immediate survival
* Has received any formula feeding prior to randomization

Max Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Time to full enteral feeding | From the start of intervention until discharge home or reach a postconceptional age of 37 weeks, whichever comes first
  Full feeding volume is defined as the first day a participant receives 120 ml/kg/d for a consecutive period of 72 hours.

SECONDARY OUTCOMES:
Combined incidence of severe neonatal infections (NEC, LOS, Meningitis) and mortality | From the start of intervention until discharge home or reach a postconceptional age of 37 weeks, whichever comes first
  LOS: defined as one positive bacterial culture in blood occurring > 3 days after birth with clinical signs of infection and with antibiotics treatment for ≥ 5 days.
  Clinical sepsis: Negative bacterial culture in blood, but the infants have clinical signs of infection and fulfil more than 2 of the following criteria: (1) Decrease in WBC , or increase in WBC(2) Immature//total neutrophils ≥0.16; (3) CRP ≥8 μg/mL; (4) Procalcitonin ≥ 2 ng/mL; (5) Platelets ≤ 100 ×109/ L.
  Meningitis: Positive bacterial culture from cerebrospinal fluid (CSF) with clinical signs. When negative, if the infants have clinical signs of meningitis and have the following changes in leucocyte counts or biochemistry values in CSF: 1) increase in leucocytes, 2) increase in total protein, and 3) increase in glucose, clinical meningitis should be recorded.
  NEC: Stage II or III according to modified Bell's criteria
The presence of feeding intolerance | From the start of intervention until discharge home or reach a postconceptional age of 37 weeks, whichever comes first
  Presence of feeding intolerance is defined as at any time when feeding is withheld by the neonatologists from day 1-7 and from day 8-14. The number of withheld meals of the prescribed feeding volume, and actually received volume from day 1-7 and from day 8-14, are recorded to indicate the degree of feeding intolerance.
Volume and color of gastric residual | From the start of intervention until discharge home or reach a postconceptional age of 37 weeks, whichever comes first
  The volume and color of gastric residuals withdrawn from the gastric tube are recorded by attending nurses, prior to a feeding
Days on PN | From the start of intervention until discharge home or reach a postconceptional age of 37 weeks, whichever comes first
  Days on PN are the total number of days that a participant receives any i.v. protein and/or lipid.
Days to regain birth weight | From the start of intervention until discharge home or reach a postconceptional age of 37 weeks, whichever comes first
  Days to regain birth weight is the total number of days that an infant used to regain his/her birth weight
Days of hospitalization | From the start of intervention until discharge home or reach a postconceptional age of 37 weeks, whichever comes first
  Total number of days that a participant is hospitalized in the neonatal department for
Body weight, length, and head circumference | Weekly until discharge home or reach a postconceptional age of 37 weeks, whichever comes first
  The weight, length, and head circumference of participants are measured every week
Blood tests on day 7 and 14 (extracted from patient charts) | Postnatal day 7 and 14
  Blood tests are performed according to the standard practices at each hospital, including blood gas, hematology, CRP, blood biochemistry for liver and kidney functions, bone health (e.g. phosphate and bone-specific alkaline phosphatase), mineral status (including sodium, potassium, calcium, chloride, and phosphate), blood lipid profile, and blood glucose.

CONTACTS AND LOCATIONS:
Overall Officials: Per Sangild, PhD, Study Chair — University of Copenhagen
Locations (8):
- China (8):
  - Dongguan Women and Children's Hospital, Dongguan, Guangdong
  - Foshan Maternal and Child Health Hospital, Foshan, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Longgang District Central Hospital of Shenzhen, Shenzhen, Guangdong
  - Shenzhen Luohu Maternal and Child Health Hospital, Shenzhen, Guangdong
  - Shenzhen Nanshan Maternal and Child Health Hospital, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - University of Chinese Academy of Sciences-Shenzhen Hospital, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yan X, Pan X, Ding L, Dai Y, Chen J, Yang Y, Li Y, Hao H, Qiu H, Ye Z, Shen RL, Li Y, Ritz C, Peng Y, Zhou P, Gao F, Jiang PP, Lin HC, Zachariassen G, Sangild PT, Wu B. Bovine colostrum to supplement the first feeding of very preterm infants: The PreColos randomized controlled trial. Clin Nutr. 2023 Aug;42(8):1408-1417. doi: 10.1016/j.clnu.2023.06.024. Epub 2023 Jun 28. PMID 37437359
- [Derived] Juhl SM, Ye X, Zhou P, Li Y, Iyore EO, Zhang L, Jiang P, van Goudoever JB, Greisen G, Sangild PT. Bovine Colostrum for Preterm Infants in the First Days of Life: A Randomized Controlled Pilot Trial. J Pediatr Gastroenterol Nutr. 2018 Mar;66(3):471-478. doi: 10.1097/MPG.0000000000001774. PMID 29019855